CLINICAL TRIAL: NCT01779102
Title: A Phase II/III Trial Investigating if Concomitant Injections of the Diagnostic Agents C-Tb and 2 T.U Tuberculin PPD RT 23 SSI Affect the Induration Responses in Combination With a Safety Assessment of C-Tb
Brief Title: Safety Study Investigating if Concomitant Injections of C-Tb and 2 T.U Tuberculin Affect Induration Responses
Acronym: TESEC-07
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: TESEC-07
Record Dates: First submitted 2013-01-18; First posted 2013-01-30 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.1 µg C-Tb (Experimental): The C-Tb agent is given alone to volunteers in the RIGHT or LEFT forearm according to a double blind randomisation scheme
  Interventions: Biological: C-Tb
- 2 T.U Tuberculin PPD RT 23 SSI (Active Comparator): The 2 T.U Tuberculin PPD RT 23 SSI agent is given alone to volunteers in the RIGHT or LEFT forearm according to a double blind randomisation scheme
  Interventions: Biological: Tuberculin PPD RT 23 SSI
- 0.1 µg C-Tb / 2 T.U Tuberculin PPD (Experimental): The C-Tb and 2 T.U Tuberculin PPD RT 23 SSI agents are given concomitantly to volunteers in the RIGHT and LEFT forearms according to a double blind randomisation scheme
  Interventions: Biological: C-Tb / Tuberculin PPD RT 23 SSI

INTERVENTIONS:
Biological: C-Tb — C-Tb is administered by the Mantoux injection technique to each volunteer in the RIGHT or LEFT forearm according to a double blind randomisation scheme
  Arms: 0.1 µg C-Tb
Biological: Tuberculin PPD RT 23 SSI — Tuberculin is administered by the Mantoux injection technique to each volunteer in the RIGHT or LEFT forearm according to a double blind randomisation scheme
  Arms: 2 T.U Tuberculin PPD RT 23 SSI
Biological: C-Tb / Tuberculin PPD RT 23 SSI — The C-Tb and Tuberculin agents are administered by the Mantoux injection technique to each volunteer in the RIGHT and LEFT forearm according to a double blind randomisation scheme
  Arms: 0.1 µg C-Tb / 2 T.U Tuberculin PPD

SUMMARY:
A new, more specific skin test to detect tuberculosis has been developed by Statens Serum Institut in Denmark. The new skin test is named C-Tb and like the current Tuberculin a positive test result will show as redness and/or induration at the injection site, while a negative test will leave no reactions.

The aim of this study is to address if the size of induration and the sensitivity of C-Tb is influenced by concomitant injections of C-Tb and Tuberculin. Furthermore, the intention is to evaluate the safety of C-Tb when injected alone or concomitantly with Tuberculin.

DETAILED DESCRIPTION:
The TESEC-07 trial is a GCP double blind randomised controlled phase II/III trial investigating if concomitant injections of the diagnostic agents C-Tb and 2 T.U Tuberculin PPD RT 23 SSI affect the induration responses in combination with a safety assessment of C-Tb. TESEC-07 is a multi-centre trial and will be conducted in South Africa in patients recently diagnosed with TB comprising 360 HIV negative and 90 HIV positive adults allocated to 3 trial groups.

* A within group paired comparison of 0.1 μg/0.1 mL C-Tb and PPD RT 23 in 150 TB patients. The C-Tb and PPD RT 23 agents are given concomitantly to each volunteer in the RIGHT AND LEFT forearms according to a randomisation scheme.
* A group of 150 TB patients will only receive the C-Tb agent randomised to either RIGHT or LEFT forearm.
* A group of 150 TB patients will only receive the reference agent PPD RT 23 randomised to either RIGHT or LEFT forearm.

ELIGIBILITY:
Inclusion Criteria (HIV Negative patients):

* Has signed an informed consent
* Aged 18 to 65 years
* Has been diagnosed with active pulmonary TB:

  1. has a compatible clinical picture of TB according to South African guidelines with the intention to treat and 1 documented positive culture result or
  2. has a compatible clinical picture of TB according to South African Guidelines with the intention to treat and 1 documented positive GeneXpert analysis
* Is HIV negative confirmed by 2 two rapid tests
* Is willing and likely to comply with the trial procedures
* Is prepared to grant authorized persons access to their medical record

Inclusion Criteria (HIV Positive patients):

* Has signed an informed consent
* Aged 18-65 years
* Has been diagnosed with active pulmonary TB:

  1. has a compatible clinical picture of TB according to South African guidelines with the intention to treat and 1 documented positive culture result or
  2. has a compatible clinical picture of TB according to South African Guidelines with the intention to treat and 1 documented positive GeneXpert analysis
* Is HIV positive confirmed by:

  1. 2 positive rapid tests or
  2. 1 positive rapid tests and an additional confirmatory ELISA
* A CD4 count has been performed
* Is willing and likely to comply with the trial procedures
* Is prepared to grant authorized persons access to their medical records

Exclusion Criteria:

* Has been in treatment for TB for more than 2 weeks
* Has a known MDR/XDR-TB
* Has been vaccinated with a live vaccine within 6 weeks prior to the day of inclusion (e.g. MMR, yellow fever, oral typhoid vaccines) except BCG vaccine
* Has been tuberculin (TST) tested < 12 months prior to the day of inclusion
* Is pregnant, breastfeeding or intending to get pregnant
* Is a female of child bearing potential not willing to use effective barrier (including spermicidal gel), hormonal or intrauterine contraceptive measures during the trial period
* Has an active disease affecting the lymphoid organs except for HIV (e.g., Hodgkin's disease, lymphoma, leukaemia, sarcoidosis)
* Has a current skin condition which interferes with the reading of the skin tests e.g. tattoos, severe scarring, burns/sunburns, rash, eczema, psoriasis, or any other skin disease at or near the injection sites
* Has a condition where blood drawings pose more than minimal risk for the patient, such as haemophilia, other coagulation disorders, or significantly impaired venous access
* Currently participating in another clinical trial with an investigational or non investigational drug or device, or has participated in another clinical trial within the 3 months prior to dosing
* Has participated in previous clinical trials investigating the ESAT-6 and/or CFP-10 antigens
* Has a condition which in the opinion of the investigator is not suitable for participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To compare the size of induration of C-Tb and PPD RT 23 if injected alone or concomitantly in Tuberculosis infected patients (HIV positives and HIV negatives) | Onset from the injection(s) to 28 days after the injections
To assess if concomitant injections of C-Tb and PPD RT 23 influence the tests abilities to identify positive results of Tuberculosis in Tuberculosis infected patients | Onset from the injection(s) to 28 days after the injections

SECONDARY OUTCOMES:
To compare the C-Tb test's ability to identify positive results in Tuberculosis infected patients with the in vitro QuantiFERON®TB Gold In Tube assay in blood collected immediately before application of the C-Tb skin test | Onset from the injection(s) to 28 days after the injections
To compare the C-Tb test's ability to identify positive results in Tuberculosis infected patients with the PPD RT 23 test | Onset from the injection(s) to 28 days after the injections
To assess the safety of C-Tb skin test by investigating laboratory safety parameters and assessing all adverse events (local and systemic) occurring within 28 days after administration of the C-Tb and/or PPD RT 23 tests | Onset from the injection(s) to 28 days after the injections

CONTACTS AND LOCATIONS:
Overall Officials: Pernille N Tingskov, BN, RN, Study Director — Statens Serum Institut; Keertan Dheda, MD, Prof, Principal Investigator — UCT Lung Institute, University of Cape Town
Locations (7):
- South Africa (7):
  - TASK, M2, Karl Bremer Hospital,, Cape Town, Cape Town
  - Tiervlei Trial Centre, Karl Bremer Hospital, Cape Town, Cape Town
  - UCT Lung Institute, Cape Town, Cape Town
  - Primecure Medicentre, Port Elizabeth, Port Elizabeth
  - Synexus Stanza Bopape Clinic, Pretoria, Pretoria
  - Setshaba Research Centre, Pretoria, Pretoria
  - Be Part Yoluntu Centre, Paarl, Western Cape

REFERENCES:
- [Derived] Aggerbeck H, Ruhwald M, Hoff ST, Tingskov PN, Hellstrom E, Malahleha M, Siebert M, Gani M, Diacon A, Novelijc Z, Andersen P, Dheda K. Interaction between C-Tb and PPD given concomitantly in a split-body randomised controlled trial. Int J Tuberc Lung Dis. 2019 Jan 1;23(1):38-44. doi: 10.5588/ijtld.18.0137. Epub 2018 Dec 20. PMID 30572979